CLINICAL TRIAL: NCT05770583
Title: Determination of the Incidence of Hyperoxia and the Effectiveness of FiO2 Titration Guided by the Oxygen Reserve Index in Preventing Hyperoxia.
Brief Title: The Effectiveness of FiO2 Titration Guided by the Oxygen Reserve Index in Preventing Hyperoxia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aykut Saritas, associated professor, Tepecik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Tepecik Training and research
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hyperoxia; Complication
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen Saturation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Fraction of inspired oxygen (FiO2) is titrated guided by oxygen saturation in that range; %95<oxygen saturation≤%98
  Interventions: Procedure: SpO2 (oxygen saturation)
- ORi+SpO2 (oxygen saturation) group (Experimental): * FiO2 will be titrated by reducing 10% if Ori>0.01 andSpO2 ≥ 98% until Ori is 0.00.
  * FiO2 will not be changed if Ori is 0.00 and %95<oxygen saturation≤%98
  * FiO2 will be increased by 10% if oxygen saturation <95 or PaO2<60 mmHg
  Interventions: Procedure: Titration of fraction of inspired oxygen (FiO2) guided by ORI and oxygen saturation

INTERVENTIONS:
Procedure: Titration of fraction of inspired oxygen (FiO2) guided by ORI and oxygen saturation — * FiO2 will be titrated by reducing 10% if Ori>0.01 and oxygen saturation ≥ 98% until Ori is 0.00.
  * FiO2 will not be changed if Ori is 0.00 and %95<oxygen saturation≤%98
  * FiO2 will be increased by 10% if oxygen saturation <95 or PaO2<60 mmHg
  Other Names: ORİ+SpO2
  Arms: ORi+SpO2 (oxygen saturation) group
Procedure: SpO2 (oxygen saturation) — Fraction of inspired oxygen (FiO2) is titrated guided by oxygen saturation in that range; %95<oxygen saturation≤%98
  Arms: Control group

SUMMARY:
Oxygen therapy is the most common treatment modality for patients with hypoxemia, but target values for normoxemia are not clearly defined. Therefore, iatrogenic hyperoxemia is a very common situation. Even though there are many side effects reported related to hyperoxemia and hyperoxemia is shown to be related to worse outcome than expected; clinicians still observe hyperoxemia frequently.

Oxygen reserve index (ORi™) (Masimo Corp., Irvine, USA) can guide clinicians in detection of hyperoxia. ORi is a parameter which can evaluate partial pressure of oxygen (PaO2) rating from 0 to 1. There are growing evidences in ORi that it might be helpful to reduce hyperoxia in general anesthesia. Continuous ORi monitoring can be used for detecting and preventing hyperoxia. The ability to perform FiO2 titration with ORi may be an appropriate monitoring management to prevent the harmful effects of hyperoxia.In this study, in patients who underwent major abdominal surgery; It was aimed to investigate the effectiveness of ORi-guided FiO2 titration in preventing hyperoxia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18,
2. Patients scheduled for major abdominal surgery that are expected to last longer than 2 hours
3. Patients that have invasive arterial monitorization
4. American Society of Anesthesiologists physical class I, II or III.

Exclusion Criteria:

1. Patients younger than 18
2. Patients that need to be treated with high doses of vasopressors,
3. Patients having peripheric hypoperfusion,
4. Hemodynamically unstable patients,
5. Patients with hemoglobinopathy,
6. Pregnancy,
7. Morbid obesity (bmi>40 kg/m2),
8. Patients with arrythmia that can result in hemodynamic instability, patients with acute coronary syndrome
9. Acute respiratory failure or ARDS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Correlation of FiO2 and ORi value | Until the surgery is over
  Correlation of FiO2 value and ORi value. FiO2 adjusted until ORi reaches to zero and %95<oxygen saturation≤%98
Correlation of PaO2 and ORİ value | Until surgery is over
  Pressure of arterial oxygen is obtain from arterial blood gas analysis as usual practice in 10 min and every hour until surgery is over

SECONDARY OUTCOMES:
Fraction of inspired oxygen (FiO2) | First 10 th min after intubation and every hour until surgery is over
  Fraction of inspired oxygen (FiO2) administered during the surgery
Systolic blood pressure (SBP) | First 10 th min after intubation and every hour until surgery is over
  Measurement of systolic blood pressure (SBP)
Diastolic blood pressure (DBP) | First 10 th min after intubation and every hour until surgery is over
  Measurement of diastolic blood pressure (DBP)
Heart rate (HR) | First 10 th min after intubation and every hour until surgery is over
  Measurement of heart rate (HR)
Positive end-expiratory pressure (PEEP) | First 10 th min after intubation and every hour until surgery is over
  Measurement of PEEP

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Research and Training Hospital, Izmir, Konak, Turkey (Türkiye)

REFERENCES:
- [Background] Pala Cifci S, Urcan Tapan Y, Turemis Erkul B, Savran Y, Comert B. The Impact of Hyperoxia on Outcome of Patients Treated with Noninvasive Respiratory Support. Can Respir J. 2020 May 6;2020:3953280. doi: 10.1155/2020/3953280. eCollection 2020. PMID 32454913
- [Background] Mach WJ, Thimmesch AR, Pierce JT, Pierce JD. Consequences of hyperoxia and the toxicity of oxygen in the lung. Nurs Res Pract. 2011;2011:260482. doi: 10.1155/2011/260482. Epub 2011 Jun 5. PMID 21994818
- [Background] Vos JJ, Willems CH, van Amsterdam K, van den Berg JP, Spanjersberg R, Struys MMRF, Scheeren TWL. Oxygen Reserve Index: Validation of a New Variable. Anesth Analg. 2019 Aug;129(2):409-415. doi: 10.1213/ANE.0000000000003706. PMID 30138170
- [Background] Yoshida K, Isosu T, Noji Y, Ebana H, Honda J, Sanbe N, Obara S, Murakawa M. Adjustment of oxygen reserve index (ORi) to avoid excessive hyperoxia during general anesthesia. J Clin Monit Comput. 2020 Jun;34(3):509-514. doi: 10.1007/s10877-019-00341-9. Epub 2019 Jun 22. PMID 31227971
- [Background] Scheeren TWL, Belda FJ, Perel A. Correction to: The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):579-580. doi: 10.1007/s10877-018-0104-9. PMID 29445905